CLINICAL TRIAL: NCT04035304
Title: Online and Mobile Mindfulness Intervention to Reduce Distress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Owen, Psychologist, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35540
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Masking Description: Waitlist control group, which will receive same intervention 8 weeks after baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Coach Mobile App (Experimental): Participants in this condition will complete 3 assessments: initial, end of month two and end of month four. Each participant, following initial assessment will be provided with a link to download the Mindfulness Coach mobile app as well as with brief recommendations for how to use the app over the subsequent 16 weeks of the study. Mindfulness Coach is a mobile app for iPhone and Android, developed by the VA National Center for PTSD in collaboration with National Center for Telehealth and Technology (T2).
  Interventions: Other: Mindfulness Coach
- No Treatment Control Group (No Intervention): Participants in this condition will initially be provided with links to resources for Veterans with PTSD (http://ptsd.va.gov) and will be told that they will be contacted again in 8 weeks (60 days) to complete a second assessment. Each participant will then be provided with a link to download the Mindfulness Coach mobile app and with brief recommendations for how to use the app over the subsequent 8 weeks of the study (see description above). Participants will participate in a final follow up survey 8 weeks after receiving the app.

INTERVENTIONS:
Other: Mindfulness Coach — Mindfulness Coach provides 4 primary treatment components: 1) psychoeducation about PTSD and Mindfulness (e.g., "What is Mindfulness?", "Why Practice Mindfulness?", "Mindfulness for Veterans", "Benefits of Mindfulness for PTSD", "Practice Challenges with PTSD", and "PTSD Symptoms During Practice"), 2) self-monitoring tools for tracking mindfulness practice, 3) 9 audio- guided mindfulness exercises (e.g., "Mindful Breathing", "Body Scan", "Clouds in the Sky", etc.), and 4) reminders to regularly practice mindfulness exercises.
  Arms: Mindfulness Coach Mobile App

SUMMARY:
The purpose of this study is to test whether a mobile app can improve mindful awareness, attention, and psychological well-being in Veterans and cancer survivors with mild to moderate PTSD symptoms. Because many of those experiencing trauma symptoms do not receive evidence-based care for PTSD, it is important to identify effective means of delivering efficacious treatments, like mindfulness-based interventions, using technology-based channels. In the proposed study, Veterans with PTSD will be recruited using social media advertising and will be randomized to one of 2 groups: no treatment control group or Mindfulness Coach mobile app. Participants in each of the 2 groups will be asked to complete measures of mindfulness and psychological well- being at baseline (prior to randomization) and again at 8-weeks (immediately post-treatment) and 16-weeks (8 weeks after completing treatment).

DETAILED DESCRIPTION:
In brief, 200 community-dwelling veterans with significant, untreated PTSD symptoms will be randomized to one of 2 groups: a no-treatment control group for one month/30-days, followed by receiving the phone app. And a treatment group that will receive the Mobile app or Mindfulness Coach mobile phone app. Potential participants will be identified from targeted Facebook and other social media outreach efforts.

Investigators at Stanford/VAPAHCS will be responsible for recruitment of the Veteran sample. Those who view an advertisement will be directed to the study website, hosted by Stanford's Qualtrics domain, where they will be provided with information about the study, screened for eligibility, and then provided with an informed consent document. Participants will then be randomized to one of the two groups and provided with an invitation and hyperlink that either a) provides them with information about when they will next be contacted (30-days after initial assessment) (control group), or b) a link that allows them to download the study app (Mindfulness Coach) onto their smart phone. Participants in Group 1 will then be encouraged to use the Mindfulness Coach app as often or as little as they like. Outcomes will be evaluated using objective measures of engagement with the intervention, changes in self-report measures of mindful awareness, attention, and psychological well-being, and qualitative experiences (phone interview) associated with use of each intervention. Barriers to implementation and identified strategies for overcoming barriers will be catalogued over the duration of the study.

Description of Each Condition:

GROUP 1. Mindfulness Coach Mobile App (n = 100). Participants in this condition will complete 3 assessments: initial, end of month two and end of month four. Each participant, following initial assessment will be provided with a link to download the Mindfulness Coach mobile app as well as with brief recommendations for how to use the app over the subsequent 16 weeks of the study. Mindfulness Coach is a mobile app for iPhone and Android, developed by the VA National Center for PTSD in collaboration with National Center for Telehealth and Technology (T2). Mindfulness Coach has been widely downloaded and is the 2nd most popular VA app available to the general public. Mindfulness Coach provides 4 primary treatment components: 1) psychoeducation about PTSD and Mindfulness (e.g., "What is Mindfulness?", "Why Practice Mindfulness?", "Mindfulness for Veterans", "Benefits of Mindfulness for PTSD", "Practice Challenges with PTSD", and "PTSD Symptoms During Practice"), 2) self-monitoring tools for tracking mindfulness practice, 3) 9 audio- guided mindfulness exercises (e.g., "Mindful Breathing", "Body Scan", "Clouds in the Sky", etc.), and 4) reminders to regularly practice mindfulness exercises.

GROUP 2. Will serve, initially, as a No Treatment Control Group (n = 100) for 60- days (one-month). Participants in this condition will initially be provided with links to resources for Veterans with PTSD (http://ptsd.va.gov) and will be told that they will be contacted again in 8 weeks (60 days) to complete a second assessment. Each participant will then be provided with a link to download the Mindfulness Coach mobile app and with brief recommendations for how to use the app over the subsequent 8 weeks of the study (see description above). Participants will participate in a final follow up survey 8 weeks after receiving the app.

ELIGIBILITY:
Inclusion Criteria:

* PTSD Diagnosis
* Veteran Status
* Must own personal smartphone/tablet with internet connection
* English fluency

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Mindfulness Questionnaire | 8 weeks
  This is a 7-item questionnaire which asks participants to rate their ability to practice, and attitude towards mindfulness meditation practices. Mindfulness meditation in the clinical context is defined as nonjudgmental attention to present-moment experiences. Originally stemming from Buddhist tradition, it guides users to the regulation of their attention to maintain their focus on immediate experiences such as thoughts, emotions, body posture and sensations, and the ability to approach one's experiences with openness and acceptance. The minimum score on this scale is 7, maximum 35. Some items are reverse-coded, and possible responses include "Strongly disagree", "Somewhat disagree", "Neither agree nor disagree", "Somewhat agree", or "Strongly agree". Higher scores indicate an increased mindfulness practice capability, which is the better outcome. Responses are summed.
PEG Pain Scale | 8 weeks
  PEG is a 3-item questionnaire assessing Pain Intensity and Interference. Pain is measured on a 0 to 10 scale by asking participants to rate their pain over the past week. Responding 0 to any item indicates "No pain", whereas 10 is "Pain as bad as you can imagine". It also asks how much pain interferes with their enjoyment of life and general activity. The minimum score is 0, and maximum is 30. Lower score is the better outcome. Responses are summed.
PROMIS (Patient-Reported Outcomes Measurement Information System) Item Bank v. 1.0 - Sleep-Related Impairment - Short Form 8a | 8 weeks
  PROMIS is an 8-item questionnaire which assesses sleep quality, such as if they feel rested after sleeping, or still feel tired after they wake up, and if that impacts their quality of life. Some items are reverse-coded, and possible responses include "Not at all", "A little bit", "Somewhat", "Quite a bit", or "Very much". The minimum score is 8, and the maximum is 40. Lower score is the better outcome. Responses are summed.
Acceptance and Action Questionnaire (AAQ-II) | 8 weeks
  AAQ-II is a 10-item questionnaire on how personal memories effect feelings of anxiety and control over one's life. The Acceptance and Action Questionnaire measures experiential avoidance and psychological inflexibility, such as the avoidance of thoughts and feelings, ability to distinguish negative thoughts from objective facts about the situation, and behavioral adjustment in the presence of difficult thoughts or feelings. It is used to predict a wide-range of quality of life outcomes (e.g., depression, anxiety, general mental health, job satisfaction, future work absence, and future job performance. Some items are reverse-coded, and possible responses include "Never true", "Very seldom true", "Seldom true", "Sometimes true", "Frequently true", "Almost always true", or "Always true". The minimum score is 10, and the maximum is 70. Lower score is the better outcome. Responses are summed.
PTSD Checklist for DSM-5 (PCL-5) | 8 weeks
  The PCL-5 is a 20-item questionnaire that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including: Monitoring symptom change during and after treatment, Screening individuals for PTSD, Making a provisional PTSD diagnosis. Possible responses include "Not at all", "A little bit", "Moderately", "Quite a bit", or "Extremely". The minimum score is 0, and the maximum is 80. Lower score is the better outcome. Responses are summed.
Patient Health Questionnaire (PHQ-9) | 8 weeks
  PHQ-9 is a 10-item questionnaire that assesses the DSM-5 symptoms of Major Depression over the past two weeks. These are operationalized in the amount of impact on respondents daily functioning the symptoms have with possible responses include "Not at all", "Several days", "More than half the days", "Nearly every day". The minimum score is 0, and the maximum is 36. Lower score is the better outcome. Responses are summed.
Generalized Anxiety Disorder 7 (GAD-7) | 8 weeks
  GAD-7 is a 7-item questionnaire that assesses the DSM-5 symptoms of Generalized Anxiety Disorder symptoms over the past two weeks. These are operationalized in the amount of impact on respondents daily functioning the symptoms have with possible responses include "Not at all", "Several days", "More than half the days", "Nearly every day". The minimum score is 0, and the maximum is 28. Lower score is the better outcome. Responses are summed.
The Brief Inventory of Psychosocial Functioning (B-IPF) | 8 weeks
  B-IPF is a 7-item questionnaire that assesses posttraumatic stress disorder (PTSD)-related psychosocial functional impairment over the past month. These are operationalized in the amount of difficulty participants have in their social relationships because of their PTSD symptoms. Possible responses include "0 Not at all", "1", "2", "3 Somewhat", "4", "5", "6 Always", or "N/A". The minimum score is 0, and the maximum is 42. Lower score is the better outcome. Responses are summed.
World Health Organization Quality of Life, abbreviated version (WHOQOL) - BREF | 8 weeks
  WHOQOL - BREF is a 27-item questionnaire that assesses overall quality of life across 4 subscales over the past two weeks. The first is Physical Health, such as Activities of daily living, Dependence on medicinal substances and medical aids. Second is Psychological, such as Bodily image and appearance, memory and concentration. Third is Social relationships, such as Social support and Sexual activity. And fourth is Environment, such as Financial Resources and Physical safety and security. These subgroups are analyzed separately and not summed. Possible responses include "Very dissatisfied", "Dissatisfied", "Neither satisfied nor dissatisfied", "Satisfied", and "Very satisfied" or "Not at all", "A little", "Moderately", "Mostly", "Completely". Some items are reverse-coded. The minimum score is 27, and the maximum is 135. Higher score is the better outcome. Responses are summed.
White Bear Suppression Inventory (WBSI) | 8 weeks
  WBSI is a 15-item questionnaire that is designed to measure thought suppression. Chronic thoughts suppression is a variable that is related to obsessive thinking and negative affect associated with depression and anxiety. The WBSI can help to identify individuals who are more prone to develop chronic thought suppression as well as individuals who express wishing they were not depressed, but are in fact depressed.
  Possible responses include "Strongly disagree", "Disagree", "Neutral or don't know", "Agree", and "Strongly agree". The minimum score is 15, and the maximum is 75. Lower score is the better outcome. Responses are summed.
Five Facet Mindfulness Questionnaire | 8 weeks
  Five Facet Mindfulness is a 39-item questionnaire which assesses the participant's awareness of their thoughts, emotions, and physical state at the current moment and in general. The five facets are observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. These subgroups can be analyzed separately or summed. Possible responses include "never or very rarely true", "rarely true", "sometimes true", "often true", or "often true or always true". Some items are reverse-coded. The minimum score is 39, and the maximum is 195. Lower score is the better outcome. Responses are summed.
Multidimensional Assessment of Interoceptive Awareness (MAIA) | 8 weeks
  Multidimensional Assessment of Interoceptive Awareness is a 32-item questionnaire, of which 17 were selected, which assesses the participant's bodily awareness. It allows a more differentiated assessment of essential psychological aspects of the perception and evaluation of body sensations. The four subscales evaluated are Noticing, Not-Distracting, Not-Worrying, and Attention Regulation. Possible responses include "0 Never", "1", "2", "3", "4" or "5 Always". Higher total scores and subscale scores indicate higher levels of positive awareness, the better outcome. The minimum score is 0, and the maximum is 85. Some items are reverse coded, and subscales are averaged separately, then summed.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System Menlo Park Division, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wielgosz J, Walser RD, Kuhn E, Chang A, Bantum EO, Pagano I, Jaworski BK, Taylor K, Ramsey KM, Owen JE. Clinical benefits of self-guided mindfulness coach mobile app use for veterans with posttraumatic stress disorder: A pilot randomized control trial. Psychol Trauma. 2025 Jul;17(5):1117-1126. doi: 10.1037/tra0001736. Epub 2024 Aug 26. PMID 39190441

DOCUMENTS (1):
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT04035304/ICF_000.pdf